CLINICAL TRIAL: NCT01900964
Title: Ridge Preservation Comparing the Clinical and Histologic Healing of a PTFE Non-resorbable vs. a Collagen Membrane With an Intrasocket Mineralized Cancellous Allograft Plus a Facial Overlay Bovine Xenograft.
Brief Title: Ridge Preservation Comparing a PTFE Nonresorbable Membrane to a Collagen Membrane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Henry Greenwell, Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12.0455
Record Dates: First submitted 2013-07-10; First posted 2013-07-17 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2014-05

CONDITIONS: Clinical Efficacy
Keywords: Regeneration; Bone regeneration; Grafting, Bone; Allograft; Xenograft

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PTFE membrane (Active Comparator): A non-resorbable PTFE (polytetrafluoroethylene) membrane will be used as a positive control treatment.
  Interventions: Procedure: PTFE membrane
- Collagen membrane (Experimental): A resorbable collagen membrane will be used in the test group.
  Interventions: Procedure: Collagen membrane

INTERVENTIONS:
Procedure: PTFE membrane — The non-resorbable PTFE barrier membrane will be surgically placed in conjunction with a ridge preservation procedure.
  Arms: PTFE membrane
Procedure: Collagen membrane — A resorbable collagen membrane is surgically placed in conjunction with a ridge preservation procedure.
  Arms: Collagen membrane

SUMMARY:
A non-resorbable PTFE (teflon) membrane will be compared to a resorbable collagen membrane when used for a post-extraction ridge preservation procedure to prevent the bone loss that typically occurs. The hypothesis is that there will be no difference in the clinical and histologic results between the two membranes.

DETAILED DESCRIPTION:
Patient Selection 30 patients will be selected that meet the following criteria:

Inclusion Criteria

1. Have one non-molar tooth requiring extraction that will be replaced by a dental implant. The site must be bordered by at least one tooth.
2. Healthy male or female who is at least 18 years old.
3. Patients must sign an informed consent approved by the University of Louisville Human Studies Committee.

Exclusion Criteria

1. Patients with debilitating systemic diseases, or diseases that have a clinically significant effect on the periodontium.
2. Presence or history of osteonecrosis of jaws.
3. Patients who are currently taking IV bisphosphonates or who had IV treatment with bisphosphonates irrespective of duration.
4. Patients who have been treated with oral bisphosphonates for more than three years.
5. Patients with an allergy to any material or medication used in the study.
6. Patients who need prophylactic antibiotics.
7. Previous head and neck radiation therapy.
8. Chemotherapy in the previous 12 months.
9. Patients on long term NSAID or steroid therapy.
10. Pregnant patients.

ELIGIBILITY:
Inclusion Criteria:

1. Have one non-molar tooth requiring extraction that will be replaced by a dental implant. The site must be bordered by at least one tooth.
2. Healthy male or female who is at least 18 years old.
3. Patients must sign an informed consent approved by the University of Louisville Human Studies Committee.

   -

Exclusion Criteria:

1. Patients with debilitating systemic diseases, or diseases that have a clinically significant effect on the periodontium.
2. Presence or history of osteonecrosis of jaws.
3. Patients who are currently taking IV bisphosphonates or who had IV treatment with bisphosphonates irrespective of duration.
4. Patients who have been treated with oral bisphosphonates for more than three years.
5. Patients with an allergy to any material or medication used in the study.
6. Patients who need prophylactic antibiotics.
7. Previous head and neck radiation therapy.
8. Chemotherapy in the previous 12 months.
9. Patients on long term NSAID (nonsteroidal anti-inflammatory drug) or steroid therapy.
10. Pregnant patients. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Crestal ridge width | Time 4 months
  The crestal ridge width will be measured with a digital caliper at the baseline exam and at the 4 month examination.

SECONDARY OUTCOMES:
Percent vital bone | Time 4 months
  A trephine core will be taken at 4 months immediately prior to implant placement from the implant osteotomy site.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Greenwell, DMD, Principal Investigator — University of Louisville
Locations (1):
- Graduate Periodontics Clinic, University of Louisville, Louisvile, Kentucky, United States